CLINICAL TRIAL: NCT04009902
Title: Evaluation of Depression and Sleep Disorders in Endometriosis Patients Preoperatively and Postoperatively
Brief Title: Evaluation of Depression and Sleep Disorders in Endometriosis Patients
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.03.77
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Endometriosis; Sleep; Depression
MeSH Terms: conditions — Endometriosis; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Beck Depression Scale and Pittsburgh Sleep Quality Index — postoperative depression and sleep disorders in patients with endometriosis will be evaluated

SUMMARY:
The aim of this study was to compare the depression and sleep disturbances of operated endometriosis patients before and after the operation. The main objective here is to provide data on how patients' psychological states and sleep patterns are affected by the symptoms of endometriosis and how these effects can be corrected. In this way, it is aimed to determine whether the patients have psychological support needs and to give the planned treatment due to endometriosis in the early period. As a secondary goal, it is planned to keep the patients in follow-up with their improved sleep and psychological conditions, and to improve their adherence to treatment and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years of age with no known psychiatric disorder and
* Endometriosis patients with indications for operation

Exclusion Criteria:

* Patients receiving only medical treatment without any indication for operation,
* those with a known psychiatric disease,
* patients with sleep disorders due to another reason,
* Patients over the age of 49, patients under the age of 18,
* Patients with malignancy,
* pregnant women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study group included patients with indications for operation and who agreed to test for depression and sleep disorders.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
Beck Depression Scale | 1 week
  postoperative depression in endometriosis patients will be evaluated. Consists of 21 questions scored between 0-3.
  HIGH SCORE SHOWS TO HIGH DEPRESSION. (0-63 POINTS)
Pittsburgh Sleep Quality Index | 1 week
  postoperative sleep disorders of endometriosis patients will be evaluated. Consists of 9 questions scored between 0-3.
  HIGH SCORE SHOWS BAD SLEEP QUALITY. (0-27 POINTS)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kanuni Sultan Süleyman Training and Research Hospital, Istanbul
  - Pınar Kadiroğulları, Istanbul